CLINICAL TRIAL: NCT04251689
Title: The Effect of Intravenous Mannitol Plus Saline on the Prevention of Cisplatin-induced Nephrotoxicity: A Randomized, Double-blind, Placebo Controlled Trial
Acronym: MACIN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R023h/62
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Cis-Platinum Nephropathy; Mannitol Adverse Reaction
MeSH Terms: interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): mannitol 20 gram plus 0.9% normal saline 100 ml one hour after cisplatin
  Interventions: Drug: Mannitol
- placebo (Placebo Comparator): 0.9% normal saline 100 ml one hour after cisplatin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mannitol — Mannitol 20 gram plus 0.9% normal saline 100 ml one hour after cisplatin
  Arms: intervention
Drug: Placebo — 0.9% normal saline 100 ml
  Arms: placebo

SUMMARY:
This study include cancer patients who had received chemotherapy that include cisplatin. Patients were randomly assigned to either a mannitol 20 g intravenous single dose after cisplatin or a placebo (saline). The primary outcome was to compare acute kidney injury (AKI), which was defined as increase creatinine 0.3 mg/dl in 48 hours by KDIGO criteria using serum creatinine and 24 hour urine creatinine to calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who was at least 18 years old.
2. Patients who had been diagnosed with cancer proven by tissue biopsy.
3. Patients who were scheduled to receive cisplatin or combination of cisplatin and other chemotherapy, which the dose of cisplatin was not exceeded 100 mg/m2.
4. Patients were required to have a normal renal function (GFR > 60 mL/min/1.73m2).
5. Patients with an Eastern Cooperative Oncology Group (ECOG) score ≤ 2.
6. Patients with normal serum sodium and serum potassium level.

Exclusion Criteria:

1. Patients with any acute kidney injury event before randomized into trial not more than 6 months.
2. Patients with chronic kidney disease or hydronephrosis.
3. Patients with history of nephrectomy.
4. Patients who had previously received immunosuppressants for any immune deficiency disease.
5. Patients with who had received chemotherapy which induce nephrotoxicity.
6. Patients with had received drug which is nephrotoxic (amphotericin B, aminoglycoside or non-steroidal anti-inflammatory drug).
7. Patients who had cirrhosis with child pugh score more than 7.
8. Patients with or had a known allergy to cisplatin or mannitol.
9. Patients with chronic heart failure who cannot received fluid more than 1 liter.
10. Patients who were not comfortable to follow up at clinic for long term outcome.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-02-14 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | 48 hours
  Rate of patients with serum creatinine increase 0.3 mg/dl or ≥50% or urine output of <0.5 mL/kg/hour for >6 hours by AKIN criteria

SECONDARY OUTCOMES:
Decline 24-hour urine creatinine clearance | 48 hours
  Rate of patients with lower than 60 mL/min/1.73m2 of 24-hour urine creatinine clearance after receiving cisplatin

CONTACTS AND LOCATIONS:
Locations (1):
- Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided